CLINICAL TRIAL: NCT07155005
Title: Evaluating the Safety and Effectiveness of Steerable Ureteroscopic Renal Evacuation (SURE) With the CVAC® System Compared to Other Therapeutic Interventions for the Treatment of Renal Stones: a Prospective, Observational Trial
Brief Title: Stone Clearance With Aspiration vs Other Technologies: a Real-world Evidence Study
Acronym: SCORE
Status: Not yet recruiting | Type: Observational
Sponsor: Calyxo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP00007
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Urolithiasis; Stones, Kidney; Renal Stones; Kidney Stones
Keywords: ureteroscopy; CVAC; SURE; URS
MeSH Terms: conditions — Urolithiasis; Kidney Calculi; Nephrolithiasis | interventions — Ureteroscopy; Dust; Nephrolithotomy, Percutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (5):
- PERCUTANEOUS NEPHROLITHOTOMY (PCNL): This is a surgical procedure under general anesthesia, where a rigid probe is placed through the flank, creating a percutaneous tract into the renal collecting system under fluoroscopy. Via nephoscopy, stones are fragmented, pulverized, and extracted.
  Interventions: Procedure: PERCUTANEOUS NEPHROLITHOTOMY (PCNL)
- DIRECT IN-SCOPE SUCTION (DISS) IN FLEXIBLE URETEROSCOPY (FURS): DISS is a system that integrates controlled suction into the working channel of a standard flexible ureteroscope during ureteroscopic lithotripsy. A suction adapter is attached externally to the ureteroscope's working port, which connects to a standard hospital suction source.
  Interventions: Device: DIRECT IN-SCOPE SUCTION (DISS) IN FLEXIBLE URETEROSCOPY (FURS)
- URETEROSCOPY (URS) WITHOUT SUCTION: URS allows the surgeon to visualize the stone by inserting the ureteroscope into the ureter, most often a flexible scope that allows them to accommodate to the shape of the ureter and renal collecting system. A laser fiber is advanced through the working channel of the ureteroscope to perform stone fragmentation (dusting or breaking up the calculi). Once the stones are dusted or fragmented, the pieces can be removed by active extraction of individual stone fragments using a retrieval basket or using the concept of stone dusting where the fragments are small enough to be passed after the procedure.
  Interventions: Procedure: URETEROSCOPY (URS) WITHOUT SUCTION
- FLEXIBLE AND NAVIGATIONAL URETERAL ACCESS SHEATH (FANS) IN FLEXIBLE URETEROSCOPY (FURS): FANS is designed to incorporate suction to facilitate stone fragment removal through its lumen and is used with a separate ureteroscope. FANS is fitted with a Y connector with a pressure control vent and connects to a standard vacuum device. A separate ureteroscope provides direct visualization and irrigation and a separate specimen collector captures stone debris.
  Interventions: Device: FLEXIBLE AND NAVIGATIONAL URETERAL ACCESS SHEATH (FANS) IN FLEXIBLE URETEROSCOPY (FURS)
- CVAC® SYSTEM: The CVAC Aspiration System is a sterile, single use, steerable ureteral catheter system with integrated vision, irrigation and aspiration for the treatment and removal of urinary stones (kidney stones, fragments, and dust).
  Interventions: Device: CVAC® SYSTEM

INTERVENTIONS:
Device: CVAC® SYSTEM — The CVAC Aspiration System is a sterile, single use, steerable ureteral catheter system with integrated vision, irrigation and aspiration for the treatment and removal of urinary stones (kidney stones, fragments, and dust).
  Other Names: SURE; CVAC
  Groups: CVAC® SYSTEM
Device: FLEXIBLE AND NAVIGATIONAL URETERAL ACCESS SHEATH (FANS) IN FLEXIBLE URETEROSCOPY (FURS) — Group/Cohort Description: FANS is designed to incorporate suction to facilitate stone fragment removal through its lumen and is used with a separate ureteroscope. FANS is fitted with a Y connector with a pressure control vent and connects to a standard vacuum device. A separate ureteroscope provides direct visualization and irrigation and a separate specimen collector captures stone debris.
  Other Names: FANS
  Groups: FLEXIBLE AND NAVIGATIONAL URETERAL ACCESS SHEATH (FANS) IN FLEXIBLE URETEROSCOPY (FURS)
Device: DIRECT IN-SCOPE SUCTION (DISS) IN FLEXIBLE URETEROSCOPY (FURS) — DISS is a system that integrates controlled suction into the working channel of a standard flexible ureteroscope during ureteroscopic lithotripsy. A suction adapter is attached externally to the ureteroscope's working port, which connects to a standard hospital suction source.
  Other Names: DISS
  Groups: DIRECT IN-SCOPE SUCTION (DISS) IN FLEXIBLE URETEROSCOPY (FURS)
Procedure: URETEROSCOPY (URS) WITHOUT SUCTION — URS allows the surgeon to visualize the stone by inserting the ureteroscope into the ureter, most often a flexible scope that allows them to accommodate to the shape of the ureter and renal collecting system. A laser fiber is advanced through the working channel of the ureteroscope to perform stone fragmentation (dusting or breaking up the calculi). Once the stones are dusted or fragmented, the pieces can be removed by active extraction of individual stone fragments using a retrieval basket or using the concept of stone dusting where the fragments are small enough to be passed after the procedure.
  Other Names: URS; Dusting; Basketing
  Groups: URETEROSCOPY (URS) WITHOUT SUCTION
Procedure: PERCUTANEOUS NEPHROLITHOTOMY (PCNL) — This is a surgical procedure under general anesthesia, where a rigid probe is placed through the flank, creating a percutaneous tract into the renal collecting system under fluoroscopy. Via nephoscopy, stones are fragmented, pulverized, and extracted.
  Other Names: PCNL
  Groups: PERCUTANEOUS NEPHROLITHOTOMY (PCNL)

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of SURE with the CVAC System compared to other therapeutic interventions for the removal of renal stones in subjects that are candidates for URS with laser lithotripsy.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for ureteroscopy with laser lithotripsy
* Be willing and able to return for and respond to all study-related follow up procedures
* Have been informed of the nature of the study and has provided informed consent using the IRB approved informed consent (ICF)

Exclusion Criteria:

* Untreated urinary tract infection at the time of the index procedure
* Significant comorbidities
* Bladder, ureteral or kidney abnormalities
* Pregnant individuals
* Unable to meet the treatment and follow up protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidate for ureteroscopy with laser lithotripsy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Residual Stone Volume (RSV) | 30-Day